CLINICAL TRIAL: NCT04083573
Title: Comparison of Diagnostic Performance of Medical Monitor and Medical Augmented Reality Glasses in Endoscopy: Observation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Chan Gyoo Kim, Senior Scientist, National Cancer Center, Korea
Other Study IDs: NCC2019-0153
Record Dates: First submitted 2019-08-26; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: application of medical augmented reality glasses — Endoscopic images from medical monitor and medical augmented reality glasses will be collected and reviewed. Outcomes from both series of images will be compared

SUMMARY:
The purpose of this study was to compare the outcomes of medical augmented reality glasses and general monitors when distinguishing mucosal lesions from submucosal lesions in endoscopic diagnosis for early gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early gastric cancer who are scheduled for endoscopic submucosal dissection
* Age 19 or more
* Patients who voluntarily participated in this clinical study and signed a written informed consent

Exclusion Criteria:

* Patients with poor general medical condition which does not allow them to understand and submit a informed consent
* Patients who do not agree with this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early gastric cancer who are scheduled for endoscopic submucosal dissection will be the study population
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Consistency between the result from medical monitor and that from medical augmented reality glass | Image review will be conducted after full collection of both series of images. Review process will be done within 3 months after acquision of images. The time for study completion is aimed at 1 year from the start date.
  All series of images will be reviewed by several endoscopists by evaluation of several endoscopic findings.
  Then, concordance rate between the result from medical monitor and that from medical augmented reality glass will be assessed.
  More specifically, % of patients that does not show the same results (m cancer, sm cancer, or indeterminate) between medical monitor and medical augmented reality will be assessed.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoon JW, Chen RE, Kim EJ, Akinduro OO, Kerezoudis P, Han PK, Si P, Freeman WD, Diaz RJ, Komotar RJ, Pirris SM, Brown BL, Bydon M, Wang MY, Wharen RE Jr, Quinones-Hinojosa A. Augmented reality for the surgeon: Systematic review. Int J Med Robot. 2018 Aug;14(4):e1914. doi: 10.1002/rcs.1914. Epub 2018 Apr 30. PMID 29708640
- [Background] Takeshita H, Kihara K, Yoshida S, Higuchi S, Ito M, Nakanishi Y, Kijima T, Ishioka J, Matsuoka Y, Numao N, Saito K, Fujii Y. Clinical application of a modern high-definition head-mounted display in sonography. J Ultrasound Med. 2014 Aug;33(8):1499-504. doi: 10.7863/ultra.33.8.1499. PMID 25063416
- [Background] Eckardt C, Paulo EB. HEADS-UP SURGERY FOR VITREORETINAL PROCEDURES: An Experimental and Clinical Study. Retina. 2016 Jan;36(1):137-47. doi: 10.1097/IAE.0000000000000689. PMID 26200516
- [Background] Choi J, Kim SG, Im JP, Kim JS, Jung HC, Song IS. Endoscopic prediction of tumor invasion depth in early gastric cancer. Gastrointest Endosc. 2011 May;73(5):917-27. doi: 10.1016/j.gie.2010.11.053. Epub 2011 Feb 11. PMID 21316050